CLINICAL TRIAL: NCT01293682
Title: A Pilot Study of the Effects of High-Dose Oral Calcitriol in Breast Cancer Patients Prior to Surgery
Brief Title: Effects of High Dose Calcitriol in Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Luke Peppone, Assistant Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 25741
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Results first posted 2020-02-07 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Calcitriol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Calcitriol (Experimental): Calcitriol 45mcg/week
  Interventions: Drug: Calcitriol

INTERVENTIONS:
Drug: Calcitriol — In pill form, 45 micrograms once a week for 12 weeks
  Other Names: Rocatrol

SUMMARY:
This research will examine the effectiveness of calcitriol in treating bone loss in women who are about to begin treatment for breast cancer. Twenty-five (25) subjects are expected to take part in this study. The investigators don't know if bone loss in breast cancer survivors should be treated differently than bone loss in other women.

DETAILED DESCRIPTION:
The calcitriol intervention is aimed at reducing fracture risk by maintaining proper bone density. Calcitriol is efficacious in maintaining proper bone health and muscle mass among the general population, but little research has been done on breast cancer patients. In addition, calcitriol may be effective in reducing tumor proliferation and angiogenesis, while increasing tumor apoptosis. Each of those factors could have beneficial effects on breast cancer outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Must be female.
* Must have pathologically confirmed incident, primary invasive breast cancer.
* Must be awaiting surgical resection.
* Women of child-bearing potential (i.e. women who are pre-menopausal or not surgically sterile) must use acceptable contraceptive methods (abstinence, intrauterine device (IUD), or double barrier device) and must have a negative serum or urine pregnancy test within 1 week prior to beginning treatment on this trial. Contraceptive use needs to be continued at least 1 month after the trial has ended.
* Must provide informed consent.
* Must be willing to discontinue use of calcium and/or vitamin D supplements other than multivitamin supplementation.
* Participants must have an ionized serum calcium level within normal limits (1.19-1.29mmol/L) and a total corrected serum calcium of < 10.2mg/dl.

Exclusion Criteria:

* Subjects with life-threatening conditions that would preclude them from breast cancer treatment including: chronic cardiac failure, which is unstable despite medication use; uncontrolled hypertension; uncontrolled diabetes mellitus; or unstable coronary artery disease.
* Patients with severe metabolic disorders, which includes phenylketonuria (PKU), homocystinuria, and Fabry's disease, that would preclude them from taking calcitriol.
* Patients with a previous history of any other cancer except non-melanomous skin cancer within the past 5 years.
* Patients with impaired renal function (CRCL < 60 mL/min) or who had kidney stones (calcium salt) within the past 5 years.
* Patients with hypercalcemia (corrected serum CA > 10.2 mg/dl) or a history of hypercalcemia or vitamin D toxicity.
* Patients currently taking calcium supplements or aluminum-based antacids must immediately discontinue their use if they are to enroll in the study.
* Patients currently taking vitamin D supplements must immediately discontinue their use if they are to enroll in the study.
* Patients with a known sensitivity to calcitriol.
* Women who are pregnant or lactating.
* Women on antiresorptive drugs (e.g. bisphosphonates) within the past year.
* Women currently using oral contraception.
* Women with malabsorptive syndromes (i.e. cystic fibrosis, chronic pancreatitis) or taking medications that decrease the absorption of fat soluble vitamins (i.e. Orlistat, Questran).
* Participants assigned to calcitriol who are routinely taking a multivitamin supplement may continue the supplement as long as the amount of vitamin D in the supplement is not in excess of the RDA (recommended daily allowance) of 400 IU or 10 μg. If they are not taking a multivitamin supplement, they will be asked to not start supplementation while on study.

Ages: 18 Years to 88 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2021-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luke J Peppone, PhD, Principal Investigator — University of Rochester; Joseph J Guido, MS, Study Director — Univ of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Calcitriol
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Calcitriol
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Marital Status [Count of Participants; unit: Participants]
  Married | 7
  Divorced | 3
  Separated | 1
  Single | 1
  Widowed | 0
Education Level [Count of Participants; unit: Participants]
  Bachelor's degree or higher | 10
  Partial college training (less than 4 years) | 2
  High school graduate | 0
  Non-high school graduate | 0
Present Family Income [Count of Participants; unit: Participants]
  <$15,000 | 0
  $15,000-$29,999 | 2
  $30,000-$59,999 | 4
  >$60,000 | 5
  Unknown | 1
During the past 5 years did you regularly take a Multivitamin? [Count of Participants; unit: Participants]
  Yes | 4
  No | 8
During the past 5 years did you regularly take Vitamin D? [Count of Participants; unit: Participants]
  Yes | 4
  No | 8
During the past 5 years did you regularly take a Calcium Supplement [Count of Participants; unit: Participants]
  Yes | 5
  No | 7
Do you know or have you ever smoked 100 cigarettes in your lifetime? [Count of Participants; unit: Participants]
  Yes | 3
  No | 9

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Bone Resorption: NTX (N-terminal Telopeptide)
Description: Scale score for NTX (N-terminal telopeptide) minimum value = 4.2 nmol BCE; maximum value = 3688 nmol BCE Higher scale score for NTX indicates worse outcome.
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: nmol
Arm/Group | Calcitriol
Number analyzed (Participants) | 12
nmol | NA (NA) — The values of NTX were so low for all subjects as to be not detectable.

2. Primary Outcome: Mean Change in Bone Formation: BAP (Bone-specific Alkaline Phosphatase)
Description: Scale score for BAP (Bone-specific alkaline phosphatase) minimum value = 7 mcg/L; maximum value = 329 mcg/L Higher scale score for BAP indicates worse outcome.
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Calcitriol
Number analyzed (Participants) | 12
mcg/L | NA (NA) — The values of BAP were so low for all subjects as to be not detectable.

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Calcitriol
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 3/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Calcitriol (N=12)
Hypercalcemia (Blood and lymphatic system disorders) | 3 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-08-20): https://cdn.clinicaltrials.gov/large-docs/82/NCT01293682/Prot_SAP_000.pdf